CLINICAL TRIAL: NCT00053417
Title: Double-Blind, Placebo-Controlled, 20-Week, Parallel Group Study to Evaluate Safety, Tolerability and Activity of Oral Fampridine-SR in Subjects With Multiple Sclerosis
Brief Title: Safety and Efficacy Study of Oral Fampridine-SR in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Andrew Blight/Chief Scientific Officer, Acorda Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-F202
Record Dates: First submitted 2003-01-29; First posted 2003-01-30 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Sclerosis
Keywords: Walking Ability; Muscle strength; Spasticity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Placebo Comparator): Placebo control, twice a day (b.i.d.)
  Interventions: Drug: Placebo
- 2 (Experimental): 10 milligram (mg) fampridine b.i.d.
  Interventions: Drug: 10 milligram (mg) fampridine-SR (4-aminopyridine, 4-AP)
- 3 (Experimental): 15 mg fampridine b.i.d.
  Interventions: Drug: 15 mg fampridine-SR (4-aminopyridine, 4-AP)
- 4 (Experimental): 20 mg fampridine b.i.d.
  Interventions: Drug: 20 mg fampridine-SR (4-aminopyridine, 4-AP)

INTERVENTIONS:
Drug: Placebo — Placebo for 15 weeks
  Arms: 1
Drug: 10 milligram (mg) fampridine-SR (4-aminopyridine, 4-AP) — 2 week up titration (10 mg)
  12 weeks stable dose (10 mg)
  1 week down titration (10 mg)
  Arms: 2
Drug: 15 mg fampridine-SR (4-aminopyridine, 4-AP) — 10 mg twice daily for 1 week
  15 mg twice daily for 14 weeks
  2 week up titration (10 mg x 1 week, 15 mg x 1 week)
  12 weeks stable dose (15 mg)
  1 week down titration (10 mg)
  Arms: 3
Drug: 20 mg fampridine-SR (4-aminopyridine, 4-AP) — 2 week up titration (10 mg x 1 week, 15 mg x 1 week)
  12 weeks stable dose (20 mg)
  1 week down titration (15 mg x 3 days, 10 mg x 4 days)
  Arms: 4

SUMMARY:
Multiple Sclerosis (MS) is a disorder of the body's immune system that affects the Central Nervous System (CNS). Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the arms and legs. In people with MS, the fatty sheath that surrounds and insulates the nerve fibers (called "myelin") deteriorates, causing nerve impulses to be slowed or stopped. As a result patients with MS may experience periods of muscle weakness and other symptoms such as numbness, loss of vision, loss of coordination, paralysis, spasticity, mental and physical fatigue and a decrease in the ability to think and/or remember. These periods of illness may come (exacerbations) and go (remissions). Fampridine-SR (Sustained Release, SR) is an experimental drug that increases the ability of the nerve to conduct electrical impulses. This study will evaluate the effects of Fampridine-SR on the walking ability of subjects with MS, as well as to examine the effects on muscle strength and spasticity. The study will also examine the possible risks of taking Fampridine-SR.

ELIGIBILITY:
INCLUSION CRITERIA:

* Have a confirmed diagnosis of Multiple Sclerosis
* Are able to walk with or without an assisted device

EXCLUSION CRITERIA:

* Pregnancy, breastfeeding or females of childbearing potential not using adequate birth control
* Participating in other investigational drug trials
* A medical history or clinical findings that preclude entry into the study
* A medication history that precludes entry into the study
* Previously treated with 4-aminopyridine (4-AP)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2003-02; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (23):
  - Barrow Neurological Institute at St. Joseph Hospital and Medical Center, Phoenix, Arizona
  - USC MS Comprehensive Care Center, Los Angeles, California
  - Yale University MS Center, New Haven, Connecticut
  - Shepherd Center, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Maryland at Baltimore, Baltimore, Maryland
  - Fairview MS Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Gimbel MS Center, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Maimonides MS Care Center, Brooklyn, New York
  - Mt. Sinai School of Medicine - MS Center, New York, New York
  - University of Rochester Medical School, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Carolinas Medical Center MS Center, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health Sciences University; MS Center, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas-Houston, Houston, Texas
  - Swedish Medical MS Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- See also: Related Info — http://www.acorda.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with clinically definite MS were recruited at clinics within the US and Canada
Pre-assignment Details: 2-week placebo run-in
Groups:
- Placebo: Placebo control
- 10 mg Fampridine Twice a Day (b.i.d.): fampridine, oral, 10 mg administered twice daily
- 15 mg Fampridine b.i.d.: fampridine, oral, 15 mg administered twice daily
- 20 mg Fampridine b.i.d.: fampridine, oral, 20 mg administered twice daily
Period: Overall Study
Arm/Group | Placebo | 10 mg Fampridine Twice a Day (b.i.d.) | 15 mg Fampridine b.i.d. | 20 mg Fampridine b.i.d.
Started | 47 | 52 | 50 | 57
Completed | 45 | 50 | 49 | 51
Not Completed | 2 | 2 | 1 | 6
Not completed — Adverse Event | 1 | 0 | 1 | 5
Not completed — Non-Compliance | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Fampridine Twice a Day (b.i.d.) | 15 mg Fampridine b.i.d. | 20 mg Fampridine b.i.d. | Total
Number analyzed (Participants) | 47 | 52 | 50 | 57 | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 50 | 49 | 55 | 199
  >=65 years | 2 | 2 | 1 | 2 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 49.0 (8.99) | 49.8 (8.34) | 47.7 (8.93) | 52.2 (8.33) | 49.8 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 36 | 34 | 34 | 131
  Male | 20 | 16 | 16 | 23 | 75
Region of Enrollment [Number; unit: participants]
  United States | 42 | 47 | 45 | 51 | 185
  Canada | 5 | 5 | 5 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change From Baseline in Average Walking Speed on Timed 25-Foot Walk Test
Description: The primary efficacy variable was the percent change from baseline in average walking speed measured using the Timed 25-Foot Walk Test during the 12-week stable dose period (the average of Study Days 56, 84, and 112), relative to the mean at baseline (placebo run-in period, the average of Study Days 7 and 14).
Time Frame: Baseline (placebo run-in period); 12-week stable dose period
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | 10 mg Fampridine Twice a Day (b.i.d.) | 15 mg Fampridine b.i.d. | 20 mg Fampridine b.i.d.
Number analyzed (Participants) | 47 | 52 | 50 | 57
percent change | 1.2 (18.9) [-37.6 to 60.4] | 7.5 (22.1) [-38.9 to 103.0] | 9.7 (23.7) [-55.5 to 97.6] | 6.9 (18.5) [-40.0 to 81.4]

ADVERSE EVENTS:
Arm/Group | Placebo | 10 mg Fampridine Twice a Day (b.i.d.) | 15 mg Fampridine b.i.d. | 20 mg Fampridine b.i.d.
Serious Adverse Events (participants affected / at risk) | 2/47 | 0/52 | 4/50 | 7/57
Other Adverse Events (participants affected / at risk) | 38/47 | 45/52 | 47/50 | 52/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | 10 mg Fampridine Twice a Day (b.i.d.) (N=52) | 15 mg Fampridine b.i.d. (N=50) | 20 mg Fampridine b.i.d. (N=57)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complex Partial Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | 10 mg Fampridine Twice a Day (b.i.d.) (N=52) | 15 mg Fampridine b.i.d. (N=50) | 20 mg Fampridine b.i.d. (N=57)
Asthenia (General disorders) | 1 (1) | 10 (11) | 9 (13) | 3 (4)
Balance Disorder (Nervous system disorders) | 0 (0) | 3 (3) | 4 (4) | 5 (5)
Dizziness (Nervous system disorders) | 5 (5) | 2 (4) | 10 (14) | 7 (12)
Fall (Injury, poisoning and procedural complications) | 5 (7) | 10 (12) | 10 (23) | 5 (6)
Fatigue (General disorders) | 5 (5) | 8 (9) | 7 (10) | 5 (10)
Headache (Nervous system disorders) | 4 (4) | 6 (6) | 7 (12) | 8 (11)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5) | 10 (10) | 7 (7)
Multiple Sclerosis (Nervous system disorders) | 2 (3) | 1 (1) | 5 (5) | 5 (6)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 4 (5) | 6 (7)
Oedema Peripheral (General disorders) | 3 (4) | 4 (4) | 6 (8) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 1 (1) | 7 (13)
Paraesthesia (Nervous system disorders) | 3 (4) | 4 (4) | 3 (6) | 8 (14)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 6 (7)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 6 (8) | 5 (5) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The INSTITUTION shall submit any such manuscript or release to the SPONSOR for comment prior to publication or release at least forty-five (45) days in advance of submission for publication. If the parties disagree concerning appropriateness of the data analysis and presentation, INSTITUTION agrees to meet with SPONSOR's representatives for the purpose of making good faith efforts to discuss and resolve any issues or disagreement.